After approval by the Research Ethics Committee of the Faculty of Medical Sciences and Health of PUC-SP and filling in the terms of consent, patients were submitted to orthopedic surgery in the lower limbs, not Hospital Santa Lucinda, and eligible to participate in the study.

## Inclusion criteria:

Patients submitted to surgeries for correction of fractures in a lower hell, physical state according to an American Society of Anesthesiologists 10 I and II and age between 18 and 60 years.

## Exclusion criteria:

- (i) refusal to participate in the study;
- (ii) inability to communicate due to altered consciousness or awareness of neurological or psychiatric illness;
- (iii) contraindication to the use of non-neuraxial anesthesia or allergy to any of the drugs used without study;
- (iv) history of alcohol or drug addiction; and
- (v) history of surgery in the last 10 days.

## Drawing:

Age, sex, physical status, type of surgery, duration, history of prior surgery in the lower limbs, and presence (or not) of bladder catheterization will be recorded. Patients are randomly allocated into three groups according to a given computer-generated program measure (www.random.org):

Group D. Dexamethasone 8 mg.

Group O. Ondansetron 4 mg.

Group P. Distilled water.

For each patient, a solution to be administered through a wrap opening and sealed and containing the study group for the case. The patients involved and the data collection researchers will not be aware of the allocation. The solutions are prepared by a professional not participating in the study by diluting the agent in physiological solution or distilled water until the volume of 5 ml is complete. After a pre-anesthetic evaluation, QoR40 questionnaire and entry into the operating room, all patients are monitored with cardioscopy, noninvasive blood pressure and pulse oximetry. After a venco-lysis, midazolam will be administered intravenously before the anesthesia in titrated doses until a grade 3 or 4 sedation is obtained according to the Ramsay scale11. With the patient in position sent, the puncture subarachnoid will be performed without interspace L2-L3 or L3-L4 using 26G needle tip Quincke (B. Braun Melsungen S.A). Anesthesia will be obtained with a 0.5% hyperbaric bupivacaine injection (20 to 30 seconds) (Cristália Produtos Químicos e Farmacêuticos Ltda) at a dose of 17.5 mg if the weight is> 70 kg and / or the production> 150 minutes or 15 mg if weight <70 kg, associated with morphine (0.1 mg) without preservative (Cristália Produtos Químicos e Farmacêuticos Ltda.). The hydration will be maintained with lactated Ringer's solution. In case of failure of the block, the anesthetic procedure will be repeated or the technique will be modified for general anesthesia and the case will also be excluded. Perioperative sedation is achieved by use in metered doses (up to a maximum of 10 mg) or propofol with

the infusion rate required to achieve a level equal to or greater than 4 on a scale proposed by Ramsay.

## Post-Anesthesia Recovery Room (PACU):

Patients are referred to a PACU and will remain until a criterion is reached for a discharge (score on a modified Aldrete and Kroulik scale equal to 10). 12 During the stay in the series, in the data referring to the presence of pain, nausea, vomiting, pruritus, urinary retention, temperature below 360, length of stay and other complications. Patient without complaint of pain is evaluated every 15 minutes on the numerical scale of 0 to 10, in which "zero" means absence of pain and "ten" a stronger pain than you can imagine. Morphine 1 to 2 mg intravenously will be administered every 10 minutes for a score below 4 (1 mg for pain <7 and 2 mg for pain  $\geq$  7) when it is present. Respecting the interval of 10 minutes due to the summative effect of doses followed by morphine. However, since the patient presents with neuraxial block (spinal anesthesia), algae complaints are not expected. In view of midazolam sedation and / or proportional patient and cognitive ability to response. Nausea (and / or vomiting) treated with dimenhydrate (100mg). The pruritus will be graded according to numerical scale: zero - absence of symptoms, 1 to 3 - mild symptoms, 3 to 7 moderate modifiers and 7 to 10 - severe terms. Score above 4 will indicate the need for treatment with nalbuphine (5 mg) intravenously